CLINICAL TRIAL: NCT00002296
Title: A Multi-Center Randomized Double-Blind Placebo-Controlled Study to Investigate the Effect of Isoprinosine in Immunodepressed Patients With Uncomplicated Generalized Lymphadenopathy
Brief Title: The Safety and Effectiveness of Isoprinosine in Patients With Weakened Immune Systems and Lymph Node Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newport Pharmaceuticals International (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 008C; ISO-106-USA
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1989-06

CONDITIONS: Lymphatic Disease; HIV Infections
Keywords: T-Lymphocytes; Immune Tolerance; Inosine Pranobex; Killer Cells; T-Lymphocytes, Helper-Inducer; Acquired Immunodeficiency Syndrome; AIDS-Related Complex
MeSH Terms: conditions — Lymphatic Diseases; HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Inosine Pranobex

INTERVENTIONS:
Drug: Inosine pranobex

SUMMARY:
The objective of this Phase III, randomized, double-blind, placebo-controlled study in patients with immunologic deficiency is to determine the effect of Isoprinosine in producing an immuno-restorative response within the study observation period (including the 2-month period following cessation of the 28 days of treatment), measured by one or more of the following immunological parameters:

* Increase in natural killer (NK) cell activity.
* Increase in total T-cells (OKT-11).
* Increases in absolute number and percentage of T-helper cells (OKT-4).

ELIGIBILITY:
Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* History of gout, uric acid urolithiasis, uric acid nephrolithiasis, renal dysfunction and severe gastric ulcer.
* Lymphoid malignancy.
* Infectious mononucleosis caused by cytomegalovirus or Epstein-Barr virus.
* Heart disease (especially if receiving cardiac glycosides).
* Hemophilia.

Patients with the following are excluded:

* Kaposi's sarcoma or overt opportunistic infections as follows:
* Candida albicans, Pneumocystis carinii, Herpes simplex, Cryptococcus neoformans, Histoplasma capsulatum, Mycobacterium avium-intracellulare, Toxoplasma gondii, Legionella, Cryptosporidium, Isospora, and Papovavirus.
* Active evidence of infectious mononucleosis caused by Epstein-Barr virus (EBV) or cytomegalovirus (CMV) as determined by heterophil test (EBV) or cell culture (CMV).
* History of gout, uric acid urolithiasis, uric acid nephrolithiasis, renal dysfunction, and severe gastric ulcer.
* Critical illness.
* Condition requiring hospitalization.
* Women of childbearing age are excluded.
* Hemophilia.

Prior Medication:

Excluded:

* Steroids.
* Cytotoxic immunosuppressive agents.
* Antiviral medicine.

Prior Treatment:

Excluded:

* Radiotherapy.

Patients who have unexplained immunodepression and are at risk of developing AIDS.

* Patients with prolonged generalized lymphadenopathy for 3 or more months (greater than 1 cm at two or more noncontiguous sites).

IV drug abuse.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Newport Pharmaceuticals International Inc, Laguna Hills, California, United States